CLINICAL TRIAL: NCT00531583
Title: Autologous Peripheral Blood Stem Cell Transplantation With In Vivo Purging as an Alternate Stem Cell Transplantation Program for Pts w/AML in 1st & 2nd Complete Remission w/no HLA Matched Related Donor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC#2001-004
Record Dates: First submitted 2007-09-17; First posted 2007-09-19 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Leukemia, Monocytic, Acute
Keywords: AML in 1st & 2nd complete remission w/no HLA matched related donor
MeSH Terms: conditions — Leukemia, Monocytic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Autologous peripheral Bld Stem Cell Transplantation with In Vivo Purging as an alternate stem cell transplantation — Autologous PBSCT

SUMMARY:
Autologous peripheral Bld Stem Cell Transplantation with In Vivo Purging as an alternate stem cell transplantation program for pts w/AML in 1st & 2nd complete remission w/no HLA matched related donor

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML in 1st & 2nd complete remission w/no HLA matched related donor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2001-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Efficacy | 2009-2015

CONTACTS AND LOCATIONS:
Overall Officials: Fahad AlMohareb, Principal Investigator — KFSH&RC
Locations (1):
- KFSH&RC, Riyadh, Saudi Arabia